CLINICAL TRIAL: NCT06268002
Title: Effect of Vernonia Cinerea Lozenges as a Smoking Cessation Aid in Patients With Non-communicable Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5876557033
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2018-01

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; Vernonia Cinerea; Non-communicable disease
MeSH Terms: conditions — Smoking Cessation; Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: This study was a multicenter randomized, paralleled, double-blind, controlled trial at 5 hospitals and 2 community pharmacies in Thailand
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vernonia cinerea group (Experimental): 1 lozenges 3 times per day
  Interventions: Dietary Supplement: Vernonia cinerea
- Placebo group (Placebo Comparator): 1 placebo lozenges 3 times per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vernonia cinerea — Vernonia cinerea is an herb that is claimed in many Thai medicinal formulas. In traditional medicines, they use this herbal to treat diseases such as hypertension, asthma, fever, hepatitis, gallstones, including use to help smoker quit smoking.
  Arms: Vernonia cinerea group
Dietary Supplement: Placebo — Sweetener
  Arms: Placebo group

SUMMARY:
Vernonia cinerea is an herbal which has been recorded in many Thai herbal formulation and Thai traditional medicine has used this herbal for treating various diseases included hypertension, asthma, fever, hepatitis, kidney stone and smoking cessation. Now aday there are more interest for using Vernonia cinerea as a medication to aid smoker to quit smoking because it is cheaper than other current therapeutic medications. The objective of this study is to evaluate efficacy and safety of Vernonia cinerea lozenge for smoking cessation when compared to placebo.

DETAILED DESCRIPTION:
This study is a multicenter randomized, paralleled, double blind, controlled trial. This study will include 260 patients from Lerdsin hospital, Chest institute, Phramongkutklao hospital, Maharaj Nakorn Chiang Mai Hospital and Paolo Memorial Phaholyothin hospital who would like to quit smoke. Patients will be assigned into two groups, Vernonia cinerea group (n=130) and placebo group (n=130), both groups will be instructed to take one lozenge three times a day for three months. The two groups will receive individual counseling about smoking cessation technique by trained healthcare professional on every visit. The main primary outcome for this study is continuous abstinence rate (CAR), define as self-report of no cigarette smoking, not even a puff since target quit date, plus passed biochemical validation for 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years old
* Have at least 1 underlying non-communicable disease include hypertension, diabetes, dyslipidemia, cardiovascular diseases, cerebrovascular diseases, stable asthma (defined as no asthmatic exacerbation for the preceding 4 weeks necessitating oral prednisolone or an increased use of inhaled corticosteroid, the use of rescue treatment no more than three times a week, and with no clinical indication for change in treatment medication) COPD stage A-C according to GOLD guideline, chronic kidney diseases
* Smoke 10 cigarettes or over per day at least 1 month prior to study
* Desired to quit smoking
* Consent to participate in study

Exclusion Criteria:

* Renal dysfunction (GFR < 30 ml/mins/1.73m2)
* Liver dysfunction (Child-Pugh score C)
* Hyperkalemia (serum potassium ≥ 5 mEq/L)
* Documented of active depression or psychosis
* Active cancer
* History of acute coronary syndrome in previous 4 weeks
* Known case of pregnancy or lactation
* Use other tobacco products or other addictive substances except alcohol
* Use other smoking cessation drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
continuous abstinence rate | 1 month
  self-report of no cigarette smoking, not even a puff since target quit date, plus passed biochemical validation

SECONDARY OUTCOMES:
continuous abstinence rate (CAR) and point prevalence rate | 3,6 and 12 months
  self-report of no cigarette smoking, not even a puff since target quit date, plus passed biochemical validation

CONTACTS AND LOCATIONS:
Locations (1):
- Krittin Bunditanukul, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No